CLINICAL TRIAL: NCT03020043
Title: CardioMEMS Registry of the Frankfurt Heart Failure Center
Brief Title: Evaluation of Longterm Outcome of New York Heart Association Class III Heart Failure Patients Receiving Telemonitoring Using a Pulmonary Artery Pressure Sensor System (CardioMEMS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Birgit Assmus, PD Dr., Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Other Study IDs: FFM CardioMEMS Registry
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Invasive hemodynamic monitoring in advanced heart failure patients is a relative new option. In order to investigate the impact of remote telemonitoring of pulmonary artery pressures on mortality and morbidity in a routine clinical setting in Germany, the investigators initiated this multicenbtric registry.

DETAILED DESCRIPTION:
All patients who receive invasive hemodynamic monitoring using a pulmonary artery pressure sensor (CardioMEMS device) are offered participation in the registry. Routine heart-failure parameters, lab values, medication and QoL as obtained on the regular outpatients visits in the department are entered into a registry-specific database.

The investigators plan to asses the impact of telemonitoring on mortality, morbidity and QoL as well as on Guideline-recommended heart failure medication. In addition, it is planned to quantify the input in person time for telemonitoring.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of CardioMEMS successful
* Telemonitoring according to the SOP of the Frankfurt Heart Failure Center (Goethe University)

Exclusion Criteria:

* Unwillingness to participate in the registry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with New York Heart Association (NYHA) Class III with chronic heart failure (left and right ventricular heart failure, HFrEF, HFmrEF and HFpEF; +/- PH) , who had a hospitalisation for cardiac decompensation < 12 months
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
morbidity measured as worsening heart failure requiring hospitalisation and / or increase in diuretic dose | 5 years
  morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Assmus, MD, Principal Investigator — Klinikum Goethe University Frankfurt
Locations (2):
- Germany (2):
  - Klinikum Goethe University, Frankfurt am Main
  - University Hospital Justus-Liebe University, Giessen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herrmann E, Ecke A, Herrmann E, Eissing N, Fichtlscherer S, Zeiher AM, Assmus B. Daily non-invasive haemodynamic telemonitoring for efficacy evaluation of MitraClip(R) implantation in patients with advanced systolic heart failure. ESC Heart Fail. 2018 Oct;5(5):780-787. doi: 10.1002/ehf2.12303. Epub 2018 Jun 12. PMID 29893475
- [Result] Herrmann E, Fichtlscherer S, Hohnloser SH, Zeiher AM, Assmus B. [Implantable sensors for outpatient assessment of ventricular filling pressure in advanced heart failure : Which telemonitoring design is optimal?]. Herzschrittmacherther Elektrophysiol. 2016 Dec;27(4):371-377. doi: 10.1007/s00399-016-0472-0. Epub 2016 Nov 14. German. PMID 27844194
- [Result] Herrmann E, Ecke A, Fichtlscherer S, Zeiher AM, Assmus B. [Pulmonary artery pressure sensor for ambulatory assessment of ventricular filling pressure in advanced heart failure : What should be considered for the follow-up care?]. Herzschrittmacherther Elektrophysiol. 2018 Dec;29(4):393-400. doi: 10.1007/s00399-018-0597-4. Epub 2018 Oct 10. German. PMID 30306304